CLINICAL TRIAL: NCT04289415
Title: From Addiction to Employment. Effectiveness of Employment Support During Treatment for Substance Use Disorders. The Individual Placement and Support (IPS-SUD) Trial.
Brief Title: From Addiction to Employment.
Acronym: IPS-SUD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); Norwegian Directorate of Health (Other Government)
Responsible Party: Principal Investigator, Eline Borger Rognli, Researcher, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 54204
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Pragmatic, two-arm, parallel, superiority, randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual Placement and Support (Experimental): The intervention used in this study will be a time-limited version of IPS. The employment specialist offers up until nine months job-search support and four months in-work support, giving a total of 13 months job-related support. If a participant succeeds in obtaining work before nine months has passed the remaining job-search support months may be transferred to in-work support time.
  In the follow-up time while seeking employment, the employment specialists will work with the participants to identify skills and aspirations, establish contact with potential employers and ensure economic advice and help with benefits planning. The in-work support involves individual and regular contact with the participant and the employer.
  All participants who receive this intervention will do so in addition to their clinical treatment. The treatment provider and the employment specialist should cooperate and clarify roles together with the patient.
  Interventions: Behavioral: Individual Placement and Support
- Selv help kit and work shop (Active Comparator): The participants in the control intervention will be offered a self-help tool kit and a following introduction course to help participants see what their opportunities are, and specific tips on how to get further help. The course will last three hours a session over four days, with the offer of an individual one hour follow up session with the course leader when the course is over. The goal of the control group intervention is to enable the participants to make use of the services offered at the ordinary labor and welfare service.
  Interventions: Behavioral: Individual Placement and Support

INTERVENTIONS:
Behavioral: Individual Placement and Support — Employment specialist will work together with the participants in accordance to the method IPS in order to help the participant obtain competitive employment

SUMMARY:
Patients with substance use disorders have low employment rates and are to a large extent on the outside of the ordinary labor market. Individual Placement and Support (IPS) is an evidence based method developed to aid persons with severe mental disorders in obtaining ordinary work. IPS has been used clinically in the addiction field, but has been subject to little research. The trial "From addiction to employment" is a randomized controlled trial to investigate the effect of an IPS intervention on employment outcome among substance use disorder patients in specialized health care treatment in Oslo, Norway. The study is conducted at the Department for Substance Use Disorder Treatment at Oslo University Hospital. The trial begins to include patients March 1st 2020 and will include for two years, until February 28th 2022.

DETAILED DESCRIPTION:
The target population in this project is patients in SUD treatment who wish to gain employment. The goal of the study is to determine the effectiveness of IPS in helping persons with SUD obtain ordinary employment. A pragmatic, two-arm, parallel, superiority, randomized controlled trial will be conducted. The project is financed through innovation funding from the South Eastern Norway Regional Health Authority, the Norwegian Directorate of Health and internal resources from OUS. Participants will be allocated randomly to either an employment specialist whom they will have individual contact with for the coming 13 months or shorter (intervention), or to a self-help and four-sessions work shop intervention (control comparison). The intervention fidelity will be assessed by external evaluators according to the Norwegian translation of the IPS Fidelity Scale. Patients will be recruited to the study over a period of two years, and followed for 18 months my data collection and up until 10 years in national registries.

ELIGIBILITY:
Inclusion Criteria:

* In treatment, unemployed, want to obtain ordinary, competitive employment

Exclusion Criteria:

* coercive treatment that disables the patient to engage in the intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2032-02-28 (Estimated)

PRIMARY OUTCOMES:
Any employment | From inclusion in the trial to 18 month after inclusion in the trial
  At least 1 day of competitive employment

SECONDARY OUTCOMES:
Total time worked | From inclusion in the trial to 18 month after inclusion in the trial
  Number of days/hours worked
Time to employment | From inclusion in the trial to 18 month after inclusion in the trial
  Time from inclusion in the trial to first employment
Number of jobs | From inclusion in the trial to 18 month after inclusion in the trial
  Number of different jobs kept
Job duration | From inclusion in the trial to 18 month after inclusion in the trial
  Duration of longest employment
Employment relevant activity | From inclusion in the trial to 18 month after inclusion in the trial
  Whether the participant is engaged in education, training or other job-preparing activity
Mental distress | From inclusion in the trial and at different time points up until 12 month after inclusion in the trial
  Information obtained from the Hospital Anxiety and Depression Scale (minumum score is 0, maximum score is 42, higher score means worse outcome)
Past month substance use | From inclusion in the trial and at different time points up until 12 month after inclusion in the trial
  Information obtained from the European Addiction Severity Index
Participants' quality of life | From inclusion in the trial and at different time points up until 12 month after inclusion in the trial
  Information obtained from the EQ-5D-5L
Participants' work related quality of life | From inclusion in the trial and at different time points up until 12 month after inclusion in the trial
  Information obtained from the Work and Social Adjustment Scale (minimum score is 0, maximum score is 40, higher score means more impairment)

OTHER OUTCOMES:
Current employment status and employment during the period | From inclusion in the trial and up until 10 years after inclusion in the trial
  Information obtained from the State Register of Employers and Employees
Health Economic Cost-Benefit Assessment | From inclusion in the trial and up until 10 years after inclusion in the trial
  The assessment will include contacts with the specialized health care system (information from the National Patient Registry), contacts with the community and municipal health care and substance use treatment system (information obtained from the Municipal Patient and User Registry), reception of welfare benefits (information obtained from the FD-trygd Database) and employment (information obtained from the State Register of Employers and Employees)

CONTACTS AND LOCATIONS:
Overall Officials: Eline Rognli, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Department for Substance Use Treatment, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rognli EB, Aas EM, Drake RE, Marsden J, Anders P, Bond GR, Lystad JU, Reme SE, Arnevik EA. The effect evaluation of Individual Placement and Support (IPS) for patients with substance use disorders: study protocol for a randomized controlled trial of IPS versus enhanced self-help. Trials. 2021 Oct 15;22(1):705. doi: 10.1186/s13063-021-05673-z. PMID 34654464

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT04289415/SAP_000.pdf